CLINICAL TRIAL: NCT05892458
Title: Effect of Abdominal Massage on Prevention of Recurrent Common Bile Duct Stones After Endoscopic Sphincterotomy: A Prospective, Multicenter, Randomized Controlled Study
Brief Title: Effect of Abdominal Massage on Prevention of Recurrent Common Bile Duct Stones After Endoscopic Sphincterotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY-20232093
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Common Bile Duct Stone; Abdominal Massage
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal massage group (Experimental): The researchers demonstrated the key points of abdominal massage to patients through a video and provided a detailed explanation of the technique. Patients were encouraged to repeat and practice the massage technique after the video session. To track patient compliance, patients were required to document the frequency of their daily massages, and a designated individual collected this information via WeChat. Follow-up consultations were conducted at 1 month after enrollment and every 3 months thereafter. Patients were encouraged to contact their doctors at any time if they experienced discomfort during the study period.
  Interventions: Behavioral: Abdominal massage
- Control group (No Intervention): The control group did not receive any special intervention and were only followed up at 1 month after inclusion and every 3 months thereafter. Patients in this group were advised to contact their doctors if they experienced discomfort during the study period.

INTERVENTIONS:
Behavioral: Abdominal massage — To perform abdominal massage, patients should keep their upper body in an upright or semi-decumbent position. Using their right four fingers or palm, they should apply pressure to the middle point of the lower margin of the right upper abdominal ribs, which corresponds to the opening of the gallbladder and common bile duct. The pressure should be firm, with a depth of approximately 3-4 cm and a length of 5-10 cm, and should be applied at least once a day for 10-15 minutes per session.
  Arms: Abdominal massage group

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) and endoscopic sphincterotomy (EST) are the preferred techniques for treating common bile duct stones (CBDS) due to their advantages of minimal trauma, rapid recovery, low cost, and high success rates of up to 95%. Despite these benefits, the recurrence rate of CBDS in patients after endoscopic therapy ranges from 4% to 25%, posing a significant challenge for endoscopists and an urgent problem to be addressed.

Abdominal massage is a promising non-invasive physical intervention for preventing recurrent CBDS. This technique is a simple, effective, and non-invasive technique that can be utilized for patient self-management and is widely used in the field of digestive diseases. External pressure applied to the common bile duct during abdominal massage may promote bile excretion from the duct to the duodenum, similar to the effect of gallbladder movement flushing bile, which can prevent bile deposition in the common bile duct, thereby preventing the formation of new stones or flushing away newly-generated small stones.

Therefore, investigators plan to conduct a prospective, multicenter, randomized controlled study to investigate the preventive effect of abdominal massage in patients with recurrent CBDS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75;
* Patients with common bile duct stones recurrence;

Exclusion Criteria:

* Incomplete clearance of recurrent common bile duct stones;
* Anatomical changes (such as Billroth I/II, Roux-en-Y);
* Contraindications to abdominal massage (such as abdominal surgery, active gastrointestinal bleeding, intestinal obstruction, acute abdomen, etc.);
* Expected lifespan of less than two years;
* Unstable hemodynamics;
* Malignant arrhythmia;
* Pregnancy or lactation;
* Unwillingness or inability to sign an informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Recurrent rate of CBDS within two years | up to 2 years
  Within the two years, CBDS was found again by CT, MRCP, ERCP or biliary surgery

SECONDARY OUTCOMES:
Recurrence time of CBDS | up to 2 years
  The specific time it took for patients to have stone recurrence
Recurrence times of CBDS | up to 2 years
  The number of stone recurrences within two years
Post-ERCP complication | up to 2 years
  Adverse events after ERCP, including bleeding, perforation, biliary tract infection, and so on

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Uchida N, Hamaya S, Tatsuta M, Nakatsu T. Extracorporeal abdominal massage may help prevent recurrent bile duct stones after endoscopic sphincterotomy. Endosc Int Open. 2016 Aug;4(8):E870-3. doi: 10.1055/s-0042-109774. Epub 2016 Aug 9. PMID 27540575